CLINICAL TRIAL: NCT00080639
Title: Specialized Program Of Research Excellence (SPORE) In Ovarian Cancer/Cancer Genetics Network Collaborative Ovarian Cancer Screening Pilot Trial In High Risk Women
Brief Title: CA-125 in Screening Patients at High Risk for Ovarian Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Terminated for administrative reasons and becuase there were no enrollments
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000353332; UAB-120; UAB-0120
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Ovarian Cancer
Keywords: ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: physiologic testing
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Measuring levels of CA 125 in blood samples of women who have a high risk of developing ovarian cancer may help doctors detect cancer early and plan more effective treatment.

PURPOSE: This phase II trial is studying CA-125 levels in screening for cancer in women who are at high risk of developing ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of prospective screening for ovarian cancer in high-risk patients.
* Determine normal ranges and distributions of CA 125 within and between these patients (with subclassification by menopausal status, estrogen replacement therapy usage, and prophylactic oophorectomy).

Secondary

* Determine estimates of the specificity and positive predictive value of a risk of cancer algorithm suitable for designing a definitive trial of screening for ovarian cancer in these patients.

OUTLINE: This is a multicenter, pilot study.

Patients undergo blood collection and CA 125 levels are measured at baseline and then every 3 months for 1-2 years. Patients may be referred for an ovarian ultrasound if indicated by the CA 125 results.

Patients are followed at 6 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 2,400 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At high risk for developing ovarian cancer, as determined by meeting criteria for 1 of the following:

  * Family history of at least 2 ovarian or breast* cancers among the patient and first- and second-degree relatives within the same lineage**

    * If breast cancer* is required to meet this criterion, at least 1 breast cancer* must be premenopausal (diagnosed at age 50 or under if menopausal status unknown) NOTE: **Multiple primary cancers in the same person satisfies this criterion
  * Ashkenazi Jewish ethnicity and meets criteria for 1 of the following:

    * Prior breast cancer* diagnosis
    * One first-degree or 2 second-degree relatives with breast* or ovarian cancer

      * If breast cancer is required to meet this criterion, at least 1 breast cancer* must be premenopausal (diagnosed at age 50 or under if menopausal status unknown)
  * Probability of BRCA1 or BRCA2 mutation greater than 20%, as determined by BRCAPRO 95% posterior probability interval

    * This criterion includes the following situations for which BRCAPRO is not required:

      * Tested positive for a BRCA1 or BRCA2 mutation (100% probability)
      * First- or second-degree relative with a BRCA1 or BRCA2 mutation NOTE: *Including ductal carcinoma in situ
* No ovarian cancer, including low malignant potential cancers or primary papillary serous carcinoma of the peritoneum

PATIENT CHARACTERISTICS:

Age

* 30 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* No hemophilia
* No other bleeding disorders

Hepatic

* Not specified

Renal

* Not specified

Pulmonary

* No emphysema

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric or psychological condition that would preclude giving informed consent
* No concurrent untreated malignancy except nonmelanoma skin cancer
* No other medical condition that would preclude blood draws (e.g., chronic infectious disease)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 3 months since prior adjuvant chemotherapy for cancer

Endocrine therapy

* Concurrent adjuvant hormonal therapy (e.g., tamoxifen, leuprolide, or goserelin) allowed

Radiotherapy

* More than 3 months since prior adjuvant radiotherapy for cancer

Surgery

* More than 3 months since prior intraperitoneal surgery (laparoscopy or laparotomy)
* Prior prophylactic oophorectomy allowed

Other

* More than 5 years since prior treatment (excluding hormonal therapy) for metastatic malignancy
* No concurrent participation in other ovarian cancer early detection trials

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women know to be at high risk for ovarian cancer
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of prospective screening for ovarian cancer in high-risk patients. | baseline
Determine normal ranges and distributions of CA 125 within and between these patients (with subclassification by menopausal status, estrogen replacement therapy usage, and prophylactic oophorectomy). | baseline

SECONDARY OUTCOMES:
Determine estimates of the specificity and positive predictive value of a risk of cancer algorithm suitable for designing a definitive trial of screening for ovarian cancer in these patients. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Partridge, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama, United States